CLINICAL TRIAL: NCT01952847
Title: Randomized, Double Blinded Placebo-Controlled Study of Glutamine in Patients With Oral Mucositis on an mTOR Inhibitor-based Regimen or Esophagitis on a Regimen Receiving Radiation to the Esophagus
Brief Title: Randomized Trial of Glutamine in Patients With Mucositis or Esophagitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Per PI
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Healios Oncology Nutrition (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2013-0308; NCI-2014-00917 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-09-24; First posted 2013-09-30 (Estimated); Results first posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Mucositis; Esophagitis; mTOR Inhibitor-based Regimen; Radiation to the Esophagus; Thoracic malignancies; Placebo; Glutamine; Enterex; Glutapak-10; NutreStore; Resource; GlutaSolve; Sympt-X G.I.; Sympt-X; Questionnaires; Surveys
MeSH Terms: conditions — Mucositis; Esophagitis | interventions — Glutamine; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- mTOR Inhibitor Patient Group - Placebo (Placebo Comparator): Participants receive placebo beginning on Day 1 of an mTOR inhibitor based therapy. Placebo taken as a sugary drink by mouth. Participant will take the drink twice daily starting first day anti-cancer therapy received. Participant to swish the drink for 10 seconds and swallow. Four weeks of treatment constitute 1 cycle for participants on mTOR inhibitor therapy.
  Interventions: Other: Placebo; Behavioral: Questionnaires
- mTOR Inhibitor Patient Group - Glutamine (Experimental): Glutamine taken as a sugary drink by mouth. Participant will take the drink twice daily starting first day anti-cancer therapy received. Participant to swish the drink for 10 seconds and swallow. Four weeks of treatment constitute 1 cycle for participants on mTOR inhibitor therapy.
  Interventions: Drug: Glutamine; Behavioral: Questionnaires
- Radiation Therapy to Esophagus Patient Group - Placebo (Placebo Comparator): Placebo taken as a sugary drink by mouth. Participant will take the drink twice daily starting first day radiation therapy to the esophagus received. Participant to swallow the drink in small amounts several times.
  Interventions: Other: Placebo; Behavioral: Questionnaires
- Radiation Therapy to Esophagus Patient Group - Glutamine (Experimental): Glutamine taken as a sugary drink by mouth. Participant will take the drink twice daily starting first day radiation therapy to the esophagus received. Participant to swallow the drink in small amounts several times.
  Interventions: Drug: Glutamine; Behavioral: Questionnaires

INTERVENTIONS:
Other: Placebo — mTOR Inhibitor Patient Group: Participants receive placebo beginning on Day 1 of an mTOR inhibitor based therapy. Placebo taken as a sugary drink by mouth. Participant will take the drink twice daily starting first day anti-cancer therapy received. Participant to swish the drink for 10 seconds and swallow. Four weeks of treatment constitute 1 cycle for participants on mTOR inhibitor therapy.
  Arms: Radiation Therapy to Esophagus Patient Group - Placebo; mTOR Inhibitor Patient Group - Placebo
Drug: Glutamine — mTOR Inhibitor Patient Group - Glutamine taken as a sugary drink by mouth. Participant will take the drink twice daily starting first day anti-cancer therapy received. Participant to swish the drink for 10 seconds and swallow. Four weeks of treatment constitute 1 cycle for participants on mTOR inhibitor therapy.
  Arms: Radiation Therapy to Esophagus Patient Group - Glutamine; mTOR Inhibitor Patient Group - Glutamine
Behavioral: Questionnaires — Questionnaire completion for mTOR Inhibitor Patient Group: At baseline, Day 1 of cycle 2 and beyond, after 6 months of chemotherapy, and at end of study visit.

SUMMARY:
The goal of this clinical research study is to learn if glutamine can help control and prevent sores, blisters, or inflammation in your mouth or esophagus due to your current treatment.

In this study, glutamine will be compared to a placebo. A placebo is not a drug. It looks like the drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the flip of a coin) to 1 of 2 study groups. You will have an equal chance of being assigned to either group:

* If you are in Group 1, you will receive glutamine.
* If you are in Group 2, you will receive a placebo.

Neither you nor the study staff will know if you are receiving the study drug or the placebo. However, if needed for your safety, the study staff will be able to find out what you are receiving.

Study Drug Administration:

Glutamine or the placebo will be taken as a sugary drink by mouth. You will take the drink twice daily starting the day you first receive your anti-cancer therapy or radiation treatment.

You will mix one scoop of powder with 25-100 milliliters (about 2-6 tablespoons) of water. If you are in the chemotherapy group, you will swish the drink for 10 seconds and swallow. If you are in the radiation group, you will swallow the drink in small amounts several times.

Study Visits:

At every visit, you will be asked about any side effects you may be having and about any other drugs you may be taking.

Chemotherapy Group:

On Days 1, 8, and 22 of Cycle 1:

* You will have a mouth exam.
* Your weight will be recorded.

On Day 15 of Cycle 1:

* You will have a mouth exam.
* Your weight will be recorded.
* You will complete a quality of life questionnaire.

On Day 1 of Cycle 2 and beyond:

* You will have a mouth exam.
* Your weight will be recorded.
* If the doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for routine tests.
* You will complete a quality of life questionnaire.
* You will complete a survey about how you feel about the study drug. This should take about 5-10 minutes to complete.
* If the doctor thinks it is needed, you will have a photograph of your mouth taken.

After 3 months of chemotherapy:

* You will complete a quality of life questionnaire.

After 6 months of chemotherapy:

* Your weight will be recorded.
* You will complete a quality of life questionnaire.

Follow-Up:

For your follow-up questionnaires at Day 1 of every Cycle, at 3 and 6 months, and during the End-of-Study visit, you may be called by the study team. This call should last about 5-10 minutes.

Radiation Therapy Group:

On Weeks 1, 2, 4, and 6 of Radiation:

* You will be asked if you have inflammation of your esophagus.
* Your weight will be recorded.
* If the doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for routine tests.

On Weeks 3 and 5 of Radiation:

* You will be asked if you have inflammation of your esophagus.
* Your weight will be recorded.
* If the doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for routine tests.
* You will complete a quality of life questionnaire.
* You will complete a survey about how you feel about the study drug.

On Week 7 of Radiation:

* You will be asked if you have inflammation of your esophagus.
* Your weight will be recorded.
* If the doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for routine tests.
* You will complete a quality of life questionnaire.
* You will complete a survey about how you feel about the study drug.

  1 month after your radiation has ended:
* You will be asked if you have inflammation of your esophagus.
* Your weight will be recorded.
* If the doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for routine tests.
* You will complete a quality of life questionnaire.
* You will complete a survey about how you feel about the study drug.

  3 months after your radiation has ended:
* You will complete a quality of life questionnaire.

Follow-Up:

For your follow-up questionnaires at 1 and 3 months and during the End-of-Study visit, you may be called by the study team. This call should last about 5-10 minutes.

Length of Study:

You may continue taking the study drug for as long as the doctor thinks it is in your best interest.

You will continue taking the glutamine or placebo for 4 weeks after the completion of your anti-cancer therapy or radiation treatment. If you stop chemotherapy or radiation before completion of the intended study period, you will continue to take the study drug for 4 weeks.

If you develop severe sores, blisters, or inflammation in your mouth or esophagus, you will be removed from the study, and the doctor will give you another medication for your sores and blisters.

Your participation on the study will be over 6 months after completion of your therapy.

End-of-Study Visit:

After you are off study, you will have an end-of-study visit. For the radiation group, this will be 6 months after radiation therapy. For the chemotherapy group, this is 4 weeks after the last dose.

* Your weight will be recorded.
* If the doctor thinks it is needed, blood (about 2 teaspoons) will be drawn for routine tests.
* You will complete a quality of life questionnaire.
* If you are in the chemotherapy group, you will have a mouth exam.

This is an investigational study. Glutamine is FDA approved and commercially available for the treatment of short bowel syndrome. Its use to treat mouth sores and inflammation of the esophagus is investigational.

Up to 180 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who will be initiating therapy with any investigator-initiated mTOR inhibitor based therapy in the Department of Investigational Cancer Therapeutics (Phase I Program) or initiating radiation therapy to the esophagus.
2. For the esophagitis arm, any patient with thoracic malignancies, which will receive radiation alone or concurrent chemo/radiation. Radiation dose must be >/= 45 Gy. For the esophagitis arm, induction chemotherapy is allowed.
3. Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.
4. Patients must be >/= 17 years of age.
5. Females of childbearing potential must have a negative pregnancy test. Sexually active patients must agree to use contraception prior to, during, and 30 days after last dose.

Exclusion Criteria:

1) Patients currently receiving therapy for mucositis.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2014-07-10 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Alshawa A, Cadena AP, Stephen B, Reddy A, Mendoza TR, McQuinn L, Lawhorn K, Zarifa A, Bernhardt AM, Fessaheye S, Warneke CL, Chang JY, Naing A. Effects of glutamine for prevention of radiation-induced esophagitis: a double-blind placebo-controlled trial. Invest New Drugs. 2021 Aug;39(4):1113-1122. doi: 10.1007/s10637-021-01074-w. Epub 2021 Feb 13. PMID 33580845
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The mTOR inhibitor cohort 24 patients consented. 10 enrolled patients became ineligible after consent and before randomization due to changes in their treatment plan. The radiation cohort enrolled 53 patients; 27 were randomized to the glutamine arm and 26 were randomized to the placebo arm.
Groups:
- Radiation Therapy to Esophagus Patient Group - Glutamine: Glutamine taken as a sugary drink by mouth. Participant will take the drink twice daily starting first day radiation therapy to the esophagus received. Participant to swallow the drink in small amounts several times.
  Questionnaire completion for Radiation Therapy to Esophagus Patient Group: At baseline, Week 3, 4, 5, and 7 of radiation, and at end of study visit.
- Radiation Therapy to Esophagus Patient Group - Placebo: Placebo taken as a sugary drink by mouth. Participant will take the drink twice daily starting first day radiation therapy to the esophagus received. Participant to swallow the drink in small amounts several times.
  Questionnaire completion for Radiation Therapy to Esophagus Patient Group: At baseline, Week 3, 4, 5, and 7 of radiation, and at end of study visit.
- mTOR Inhibitor Patient Group - Placebo: Participants receive placebo beginning on Day 1 of an mTOR inhibitor based therapy. Placebo taken as a sugary drink by mouth. Participant will take the drink twice daily starting first day anti-cancer therapy received. Participant to swish the drink for 10 seconds and swallow. Four weeks of treatment constitute 1 cycle for participants on mTOR inhibitor therapy.
  Questionnaire completion for mTOR Inhibitor Patient Group: At baseline, Day 1 of cycle 2 and beyond, after 6 months of chemotherapy, and at end of study visit.
Period: Overall Study
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo
Started | 27 | 26 | 7 | 7
Completed | 25 | 24 | 7 | 6
Not Completed | 2 | 2 | 0 | 1
Not completed — Ineligible | 1 | 0 | 0 | 0
Not completed — Lack of Insurance Coverage | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Data were unavailable for 1 participant who withdrew consent after randomization but before treatment start in mTOR Inhibitor Patient Group-Placebo
Groups:
- Total: Total of all reporting groups
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo | Total
Number analyzed (Participants) | 27 | 26 | 7 | 6 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.6 (9.8) | 64.9 (11.8) | 64.3 (10.5) | 60.3 (13.4) | 65.8 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 7 | 6 | 35
  Male | 14 | 17 | 0 | 0 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 6 | 2 | 1 | 10
  White | 26 | 20 | 5 | 5 | 56
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 27 | 26 | 7 | 6 | 66
Cancer Type [Count of Participants; unit: Participants]
  Esophageal | 2 | 4 | 0 | 0 | 6
  Head & Neck | 1 | 0 | 0 | 0 | 1
  Lung | 23 | 22 | 0 | 0 | 45
  Sarcoma | 1 | 0 | 0 | 0 | 1
  Endometrial cancer | 0 | 0 | 7 | 6 | 13
BMI [Mean (Standard Deviation); unit: kg/m^2] — Height not available for mTOR cohort Population: no data for BMI taken for the mTOR cohort
  kg/m^2
    number analyzed (Participants) | 27 | 26 | 0 | 0 | 53
    (all) | 27.0 (5.1) | 28.2 (4.7) |  |  | 27.6 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Severity of Esophagitis for Radiation Therapy Patients
Description: For esophagus radiation participants, the severity of esophagitis will be taken as the highest grade observed by week six. Wilcoxon rank sum test used to compare the ordered categories of esophagitis severity.
Time Frame: 6 weeks
Population: Participants who took at least 60% of the planned doses of the study treatment and were evaluable per protocol definition.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo
Number analyzed (Participants) | 19 | 19
Participants
  Grade 1 | 2 | 0
  Grade 2 | 5 | 8
  Grade 3 | 7 | 5
  Absent | 5 | 6
Statistical Analysis 1: Comparison: Radiation Therapy to Esophagus Patient Group - Glutamine vs Radiation Therapy to Esophagus Patient Group - Placebo; Test type: Other; p = 0.73, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Severity of Oral Mucositis for mTOR Inhibitor Patients
Description: For mTOR inhibitor patients, the severity of oral mucositis will be taken as the maximum grade observed during the 6-month study period. Wilcoxon rank sum test used to compare the ordered categories of mucositis severity.
Time Frame: 6 months after start of mTOR inhibitor based treatment
Population: Evaluable Participants in the mTOR Inhibitor Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo
Number analyzed (Participants) | 7 | 6
Participants
  Grade 1 | 1 | 3
  Grade 2 | 0 | 0
  Grade 3 | 1 | 0
  Absent | 5 | 3
Statistical Analysis 1: Comparison: mTOR Inhibitor Patient Group - Glutamine vs mTOR Inhibitor Patient Group - Placebo; Test type: Other; p = 0.68, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Quality of Life (QOL) in Esophagus Radiation Patients at Baseline
Description: The Quality of Life assessed by the MD Anderson Symptom Inventory for head and neck cancer (MDASI-HN). The 13 Core symptoms include dry mouth, fatigue, pain, disturbed sleep, drowsiness, feeling of being distressed, anorexia, sadness, numbness/tingling, dyspnea, difficulty remembering, nausea, and vomiting. The 9 Head and Neck symptoms include mouth sores, problems with taste, constipation, teeth/gum problems, skin pain, difficulty with voice, choking/coughing, difficulty swallowing, and problems with mucus specific to head and neck cancers. Total symptom severity include 24 core and Head and Neck symptoms together. Symptom interference asks patients about how their symptoms impact their daily functions. The severity of each symptom and symptom interference is rated on a numerical scale from 0 (symptom is absent) to 10 (worst possible severity)." Higher scores indicate a greater symptom burden.
Time Frame: at baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo
Number analyzed (Participants) | 27 | 26
score on a scale
  Total Symptom Severity | 1.0 [0.1 to 4.0] | 1.0 [0 to 3.4]
  Core Symptom Severity | 1.4 [0.2 to 5.3] | 1.3 [0 to 4.3]
  Head & Neck symptom Severity | 0.4 [0 to 2.3] | 0.6 [0 to 3.4]
  Symptom Interference Severity | 0.5 [0 to 7.0] | 0.5 [0 to 7.2]

4. Secondary Outcome: Quality of Life (QOL) in mTOR Inhibitor Patients at Baseline
Description: as for outcome 3
Time Frame: at baseline
Measure: Median (Full Range); unit: score on a scale
Arm/Group | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo
Number analyzed (Participants) | 7 | 6
score on a scale
  Total Symptom severity | 1.0 [0.1 to 3.4] | 1.0 [0.1 to 3.9]
  Core Symptom severity | 1.3 [0.2 to 4.3] | 1.5 [0.2 to 5.0]
  Head & Neck symptom severity | 0.4 [0 to 2.6] | 0.3 [0 to 2.3]
  Symptom Interference severity | 0.3 [0 to 6.5] | 0.9 [0 to 7.7]

5. Secondary Outcome: Number of Participants With Esophagitis During 6 Weeks After Radiation Treatment Start
Description: Participants in each arm received at least 60% of planned doses of the study drug (glutamine or placebo).
Time Frame: 6 weeks
Population: Evaluable participant
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo
Number analyzed (Participants) | 19 | 19
Participants
  None | 5 | 6
  Esophagitis | 14 | 13
Statistical Analysis 1: Comparison: Radiation Therapy to Esophagus Patient Group - Glutamine vs Radiation Therapy to Esophagus Patient Group - Placebo; Test type: Superiority; p = 1.00, Fisher Exact

6. Secondary Outcome: Mucositis Incidence Per Participant During 6 Months After mTOR Inhibitor Treatment Start
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo
Number analyzed (Participants) | 7 | 6
Participants
  None | 5 | 3
  Mucositis | 2 | 3
Statistical Analysis 1: Comparison: mTOR Inhibitor Patient Group - Glutamine vs mTOR Inhibitor Patient Group - Placebo; Test type: Superiority; p = 0.59, Fisher Exact

7. Secondary Outcome: Grade 3 or Higher Esophagitis Incidence Per Participant During 6 Weeks After Radiation Start
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo
Number analyzed (Participants) | 19 | 19
Participants
  Absent, Grade 1 or 2 | 12 | 14
  Grade 3 | 7 | 5
Statistical Analysis 1: Comparison: Radiation Therapy to Esophagus Patient Group - Glutamine vs Radiation Therapy to Esophagus Patient Group - Placebo; Test type: Superiority; p = 0.73, Fisher Exact

8. Secondary Outcome: Grade 3 or Higher Mucositis Incidence Per Participant During 6 Months After Treatment Start
Time Frame: 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo
Number analyzed (Participants) | 7 | 6
Participants
  Absent, Grade 1 or 2 | 6 | 6
  Grade 3 | 1 | 0
Statistical Analysis 1: Comparison: mTOR Inhibitor Patient Group - Glutamine vs mTOR Inhibitor Patient Group - Placebo; Test type: Superiority; p = 1.00, Fisher Exact

9. Secondary Outcome: Duration of Esophagitis After Radiation Treatment Start
Time Frame: From event starts to end of study visit
Population: Participants in the radiation cohort who experienced esophagitis.
Measure: Median (Inter-Quartile Range); unit: weeks
Groups:
- Radiation Therapy to Esophagus Patient Group - Glutamine: Glutamine taken as a sugary drink by mouth. Participant will take the drink twice daily starting first day anti-cancer therapy received. Participant to swish the drink for 10 seconds and swallow. Four weeks of treatment constitute 1 cycle for participants on mTOR inhibitor therapy.
  Questionnaires: Questionnaire completion for mTOR Inhibitor Patient Group: At baseline, Day 1 of cycle 2 and beyond, after 6 months of chemotherapy, and at end of study visit.
- Radiation Therapy to Esophagus Patient Group - Placebo: Participants receive placebo beginning on Day 1 of an mTOR inhibitor based therapy. Placebo taken as a sugary drink by mouth. Participant will take the drink twice daily starting first day anti-cancer therapy received. Participant to swish the drink for 10 seconds and swallow. Four weeks of treatment constitute 1 cycle for participants on mTOR inhibitor therapy.
  Questionnaires: Questionnaire completion for mTOR Inhibitor Patient Group: At baseline, Day 1 of cycle 2 and beyond, after 6 months of chemotherapy, and at end of study visit.
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo
Number analyzed (Participants) | 14 | 13
weeks | 6.3 [1.0 to 32.4] | 7.1 [2.6 to 44.0]
Statistical Analysis 1: Comparison: Radiation Therapy to Esophagus Patient Group - Glutamine vs Radiation Therapy to Esophagus Patient Group - Placebo; Test type: Other; p = 0.54, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Duration of Mucositis After mTOR Inhibitor Treatment Start
Time Frame: From event starts to end of study visit
Population: Participants in the mTOR cohort who experienced mucositis.
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo
Number analyzed (Participants) | 2 | 3
weeks | 10.9 [6.1 to 15.7] | 9.0 [4.6 to 23.1]
Statistical Analysis 1: Comparison: mTOR Inhibitor Patient Group - Glutamine vs mTOR Inhibitor Patient Group - Placebo; Test type: Superiority; p = 1.00, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Time to Esophagitis on the Radiation Cohort Onset
Time Frame: From radiation starts to end of study visit
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo
Number analyzed (Participants) | 19 | 19
weeks | 2.9 [2.4 to 4.1] | 4.1 [3.1 to 5.9]
Statistical Analysis 1: Comparison: Radiation Therapy to Esophagus Patient Group - Glutamine vs Radiation Therapy to Esophagus Patient Group - Placebo; Test type: Superiority; p = 0.57, Log Rank

12. Secondary Outcome: Proportion of Participants Who Were Mucositis-Free at 18.3 Weeks
Description: Proportion of participants who were free of Mucositis at 18.3 weeks..
Time Frame: 18.3 weeks
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo
Number analyzed (Participants) | 7 | 6
percentage of participants | 71 [26 to 92] | 33 [1 to 75]

13. Secondary Outcome: Number of Participants With Cancer Treatment Interruptions Due to Esophagitis
Time Frame: From radiation treatment start to end of study visit, approximately 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo
Number analyzed (Participants) | 19 | 19
Participants | 0 | 0

14. Secondary Outcome: Number of Participants With Cancer Treatment Interruptions Due to Mucositis
Time Frame: 6 months after start of mTOR inhibitor based treatment
Measure: Count of Participants; unit: Participants
Arm/Group | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo
Number analyzed (Participants) | 7 | 6
Participants | 0 | 0

15. Secondary Outcome: Radiation Cohort Participant Weight Change From Baseline to End of Study
Description: Investigators recorded weight at baseline to the end of treatment with glutamine/placebo. Weight loss calculated at each study assessment visit using the Wilcoxon rank sum test.
Time Frame: from baseline to 6 months post radiation therapy
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo
Number analyzed (Participants) | 19 | 19
kg | -0.9 [-8.7 to 4.2] | -2.8 [-9.2 to 3.6]
Statistical Analysis 1: Comparison: Radiation Therapy to Esophagus Patient Group - Glutamine vs Radiation Therapy to Esophagus Patient Group - Placebo; Test type: Superiority; p = 0.83, Wilcoxon (Mann-Whitney)

16. Secondary Outcome: mTOR Inhibitor Cohort Participant Weight Change From Baseline to End of Study
Description: Investigators recorded the weight at baseline and the end of the study. Weight loss calculated at each study assessment visit using the Wilcoxon rank sum test.
Time Frame: baseline, weekly during Cycle 1, and Day 1 of Cycle 2 and beyond, and 4 weeks and 6 months after the last dose of the mTOR inhibitor
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo
Number analyzed (Participants) | 7 | 6
kg | -5.4 [-13.9 to 0.5] | -4.3 [-13.2 to -0.2]
Statistical Analysis 1: Comparison: mTOR Inhibitor Patient Group - Glutamine vs mTOR Inhibitor Patient Group - Placebo; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)

17. Secondary Outcome: Summary of Adverse Events by Grade and Relationship - Radiation Cohort
Description: CTCAE version 4.03 used to access the adverse events. Grade 1 Asymptomatic; clinical or diagnostic observations only; intervention not indicated Grade 2 Symptomatic; altered eating/swallowing; oral supplements indicated Grade 3 Severely altered eating/swallowing; tube feeding, TPN or hospitalization indicated. Total toxicity-evaluable is the total number of participants who had at least one dose of glutamine or placebo.
Time Frame: weekly during radiation, 1 month and 6 months post radiation therapy until resolution, stabilization, death, loss to follow up, or commencement of new therapy
Population: Total toxicity-evaluable is the total number of participants who had at least one dose of glutamine or placebo.
Measure: Number; unit: adverse events
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo
Number analyzed (Participants) | 25 | 24
adverse events
  Grade 3 Unlikely Related | 1 | 0
  Grade 3 Unrelated | 13 | 11
  Grade 2 Possibly related | 2 | 1
  Grade 2 Unlikely related | 0 | 0
  Grade 2 Unrelated | 15 | 15
  Grade 1 Possibly related | 3 | 0
  Grade 1 Unlikely related | 1 | 0
  Grade 1 Unrelated | 7 | 0

18. Secondary Outcome: Summary of Adverse Events by Grade and Relationship - mTOR Inhibitor Cohort
Description: as for outcome 17
Time Frame: weekly during Cycle 1, and Day 1 of Cycle 2 and beyond, and 4 weeks and 6 months after the last dose of the mTOR inhibitor until resolution, stabilization, death, loss to follow up, or commencement of new therapy
Measure: Number; unit: adverse events
Arm/Group | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo
Number analyzed (Participants) | 7 | 6
adverse events
  Grade 3 Unrelated | 3 | 3
  Grade 2 Unrelated | 0 | 2
  Grade 1 Unrelated | 6 | 6

ADVERSE EVENTS:
Time Frame: From the first dose through end of the study. Up to approximately 6 months post the radiation for the radiation therapy group. Up to 3 months, 6 months post last dose of mTOR inhibitor therapy (approximately 12 months study duration) for the mTOR inhibitor group.
Arm/Group | Radiation Therapy to Esophagus Patient Group - Glutamine | Radiation Therapy to Esophagus Patient Group - Placebo | mTOR Inhibitor Patient Group - Glutamine | mTOR Inhibitor Patient Group - Placebo
All-Cause Mortality (participants affected / at risk) | 6/25 | 2/24 | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/25 | 3/24 | 1/7 | 2/6
Other Adverse Events (participants affected / at risk) | 20/25 | 15/24 | 5/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy to Esophagus Patient Group - Glutamine (N=25) | Radiation Therapy to Esophagus Patient Group - Placebo (N=24) | mTOR Inhibitor Patient Group - Glutamine (N=7) | mTOR Inhibitor Patient Group - Placebo (N=6)
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Esophagitis (Gastrointestinal disorders) | 2 | 2 | 0 | 0
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Heart failure (Cardiac disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pulmonary hypretension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radiation Therapy to Esophagus Patient Group - Glutamine (N=25) | Radiation Therapy to Esophagus Patient Group - Placebo (N=24) | mTOR Inhibitor Patient Group - Glutamine (N=7) | mTOR Inhibitor Patient Group - Placebo (N=6)
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 17 | 13 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 3
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 5 | 3 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Odynophagia (General disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash,Maculopapular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 0 | 4 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT01952847/Prot_SAP_000.pdf